CLINICAL TRIAL: NCT06209307
Title: Preoperative Pelvic Floor Physical Therapy to Minimize Stress Urinary Incontinence After Holmium Laser Enucleation of the Prostate
Brief Title: Pelvic Floor Physical Therapy to Reduce Stress Urinary Incontinence After Holmium Laser Enucleation of the Prostate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Akhil Das, MD, FACS, Professor of Clinical Urology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3574
Record Dates: First submitted 2023-12-22; First posted 2024-01-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Hyperplasia; Stress Urinary Incontinence
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Preoperative and postoperative pelvic floor physical therapy (Experimental): Pelvic floor physical therapy (PFPT) will be initiated 1 month before surgery in patients randomized to Arm 1.
  Interventions: Behavioral: Pelvic floor physical therapy
- Arm 2: Postoperative pelvic floor physical therapy only. (No Intervention): At 1-3 days follow-up after surgery pelvic floor physical therapy (PFPT) will be initiated in the post-operative PFPT-only group as part of standard of care.

INTERVENTIONS:
Behavioral: Pelvic floor physical therapy — Pelvic floor physical therapy (i.e., Kegel exercises):
  * Finding the right muscles: To identify pelvic floor muscles, the patient should stop urination in midstream or tighten the muscles that keep from passing gas. These maneuvers use pelvic floor muscles. Once the pelvic floor muscles are identified, the patient can do the exercises in any position, although doing them lying down at first might be the easiest approach.
  * Perfecting the technique: Tighten pelvic floor muscles, hold the contraction for three seconds, and then relax for three seconds. Try it a few times in a row. When muscles get stronger, try doing Kegel exercises while sitting, standing, or walking.
  * Maintaining focus: For best results, focus on tightening only pelvic floor muscles. Be careful not to flex the muscles in the abdomen, thighs, or buttocks. Avoid breath-holding. Instead, breathe freely during the exercises.
  * Repeat 3 times a day. Aim for three sets of 10 repetitions a day.
  Arms: Arm 1: Preoperative and postoperative pelvic floor physical therapy

SUMMARY:
Holmium laser enucleation of the prostate (HoLEP) is a surgical procedure used to treat benign prostatic hyperplasia (BPH). HoLEP involves the removal of obstructive prostatic tissue via an endoscopic approach to relieve bothersome urinary symptoms. HoLEP is recommended by the American Urological Association (AUA) as a size-independent treatment for BPH. While the surgery is highly durable and versatile, post-operative stress urinary incontinence (SUI) has been reported following HoLEP, up to 44%. Pelvic floor physical therapy (PFPT) is a therapeutic strategy with low cost and risk to patients used to treat SUI following prostate surgery. However, data on the efficacy of conducting PFPT prior to HoLEP in minimizing or eliminating post-operative urinary incontinence is limited. The investigators will recruit patients who have already agreed to undergo HoLEP for this study. Participants will be randomized into two groups: The intervention group will begin standardized PFPT before surgery and will continue PFPT after surgery, and the second group will begin PFPT after surgery only (current practice). Both groups will continue with PFPT following surgery until urinary continence is regained. Investigators will compare the time required to regain urinary continence and patient-reported outcomes between the two groups.

DETAILED DESCRIPTION:
The incidence of benign prostatic hyperplasia (BPH) in men significantly increases with age and is estimated to impact over 80% of men 70 to 80 years of age. HoLEP is one of many treatments for BPH and associated lower urinary tract symptoms (LUTS). Compared to other minimally invasive surgical techniques for the treatment of BPH, HoLEP has been found to have superior outcomes and is a prostate size-independent procedure with excellent durability, high efficacy, and low complication rates. However, transient stress urinary incontinence (SUI) following HoLEP may last for several months after surgery and can lead to diminished patient quality of life (QoL) during the recovery period. Measures to prevent or reduce post-operative SUI following HoLEP, including PFPT, may improve patient outcomes.

SUI is also commonly documented after radical prostatectomy (RP) for prostate cancer. The mechanism for incontinence in both RP and HoLEP is thought to at least partially be related to temporary weakness of the external urinary sphincter, which is part of the pelvic floor musculature. While it is unclear if post-operative PFPT alone reduces SUI for patients who have undergone RP, there is evidence that PFPT started pre-operatively and continued post-operatively can decrease SUI following RP.

The utilization of pre-operative PFPT for patients undergoing HoLEP to reduce post-operative SUI is currently not well documented. To date, only one study has demonstrated evidence that PFPT prior to HoLEP may improve continence at 3 months. However, the study included patients with a BMI significantly lower than average in the United States, utilized an unclear PFPT program, and had a relatively small median prostate size (~60 mL), which is important as studies have shown that prostate size can affect post-operative incontinence.

Investigators propose a prospective randomized trial to investigate the efficacy of standardized pre-operative PFPT in reducing SUI and improving patient QoL following HoLEP. This study will help determine the role of pre-operative PFPT in the management of HoLEP-associated SUI.

ELIGIBILITY:
Inclusion Criteria:

* Adult males who have lower urinary tract symptoms (LUTS) attributed to benign prostatic hyperplasia (BPH) and considering/undergoing HoLEP for LUTS/BPH treatment at the University of California Irvine Medical Center.
* Age >= 18
* English-speaker

Exclusion Criteria:

* Non-English speaker
* Having an indwelling catheter preoperatively
* Neurological disorders that might potentially affect muscle function
* Neurogenic bladder
* Lumbosacral spine pathology
* Any condition that can interfere with pelvic muscle function per principal investigator's discretion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients will be recruited as physiologically only male patients have prostate and can develop LUTS/BPH.
Enrollment: 72 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to urinary continence following catheter removal after HoLEP | 6 months after surgery
  Time to recover from transient postoperative stress urinary incontinence

SECONDARY OUTCOMES:
Uroflow | 6 months after surgery
  Urine flow rate (milliliters/second)
Post void residual | 6 months after surgery
  Residual urine after voiding (milliliters)
American Urological Association Symptom Score | 6 months after surgery
  Validated questionnaire on urination symptoms
Operative time | Day of surgery
  Length of surgery (minutes)
Length of hospital stay | 30 days after surgery
  Days of hospitalization after surgery
Catheter duration | 30 days after surgery
  Days with catheter after surgery
Infectious complications | 30 days after surgery
  Urinary tract infection complication after surgery
Emergency room visits | 30 days after surgery
  Number of emergency room visits related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Das, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Montorsi F, Naspro R, Salonia A, Suardi N, Briganti A, Zanoni M, Valenti S, Vavassori I, Rigatti P. Holmium laser enucleation versus transurethral resection of the prostate: results from a 2-center prospective randomized trial in patients with obstructive benign prostatic hyperplasia. J Urol. 2008 May;179(5 Suppl):S87-90. doi: 10.1016/j.juro.2008.03.143. PMID 18405765
- [Background] Roehrborn CG. Benign prostatic hyperplasia: an overview. Rev Urol. 2005;7 Suppl 9(Suppl 9):S3-S14. PMID 16985902
- [Background] Michalak J, Tzou D, Funk J. HoLEP: the gold standard for the surgical management of BPH in the 21(st) Century. Am J Clin Exp Urol. 2015 Apr 25;3(1):36-42. eCollection 2015. PMID 26069886
- [Background] Das AK, Teplitsky S, Chandrasekar T, Perez T, Guo J, Leong JY, Shenot PJ. Stress Urinary Incontinence post-Holmium Laser Enucleation of the Prostate: a Single-Surgeon Experience. Int Braz J Urol. 2020 Jul-Aug;46(4):624-631. doi: 10.1590/S1677-5538.IBJU.2019.0411. PMID 32374125
- [Background] Han E, Black LK, Lavelle JP. Incontinence related to management of benign prostatic hypertrophy. Am J Geriatr Pharmacother. 2007 Dec;5(4):324-34. doi: 10.1016/j.amjopharm.2007.12.003. PMID 18179990
- [Background] Hout M, Gurayah A, Arbelaez MCS, Blachman-Braun R, Shah K, Herrmann TRW, Shah HN. Incidence and risk factors for postoperative urinary incontinence after various prostate enucleation procedures: systemic review and meta-analysis of PubMed literature from 2000 to 2021. World J Urol. 2022 Nov;40(11):2731-2745. doi: 10.1007/s00345-022-04174-1. Epub 2022 Oct 4. PMID 36194286
- [Background] Centemero A, Rigatti L, Giraudo D, Lazzeri M, Lughezzani G, Zugna D, Montorsi F, Rigatti P, Guazzoni G. Preoperative pelvic floor muscle exercise for early continence after radical prostatectomy: a randomised controlled study. Eur Urol. 2010 Jun;57(6):1039-43. doi: 10.1016/j.eururo.2010.02.028. Epub 2010 Mar 1. PMID 20227168
- [Background] Anan G, Kaiho Y, Iwamura H, Ito J, Kohada Y, Mikami J, Sato M. Preoperative pelvic floor muscle exercise for early continence after holmium laser enucleation of the prostate: a randomized controlled study. BMC Urol. 2020 Jan 23;20(1):3. doi: 10.1186/s12894-019-0570-5. PMID 31973706
- [Background] Moore KN, Cody DJ, Glazener CM. Conservative management for post prostatectomy urinary incontinence. Cochrane Database Syst Rev. 2001;(2):CD001843. doi: 10.1002/14651858.CD001843. PMID 11406013